CLINICAL TRIAL: NCT01419106
Title: SHoC-ED: Sonography in Hypotension and Cardiac Arrest in the Emergency Department.
Brief Title: Sonography in Hypotension and Cardiac Arrest in the Emergency Department.
Acronym: SHoC-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horizon Health Network (Other)
Collaborators: University of Cape Town (Other); University of Stellenbosch (Other); Dalhousie University (Other); University of Manitoba (Other); University of Saskatchewan (Other); Harvard University (Other); University of British Columbia (Other); Royal College of Emergency Medicine (Other); Canadian Association of Emergency Physicians (Industry); Saint Göran Hospital (Unknown); University of Michigan (Other)
Responsible Party: Principal Investigator, Paul Atkinson, Dr. Paul Atkinson, Professor, Department of Emergency Medicine, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2011-1590
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Hypotension; Point of Care Ultrasound; Shock
Keywords: Hypotension; Emergency care; Point of care Ultrasound; Shock
MeSH Terms: conditions — Hypotension; Shock | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): This arm of the study will NOT receive point of care ultrasound. They will receive all other standard care implemented during their visit to the ED (currently, ultrasound is NOT standard of care). The same blood tests will be done in both groups, as this will offer a means of comparing physiological changes between the two arms.
- Ultrasound (Experimental): This group WILL receive point of care ultrasound. The protocol they will receive is the ACES protocol (described above).
  Interventions: Device: Ultrasound (A point of care ultrasound protocol)

INTERVENTIONS:
Device: Ultrasound (A point of care ultrasound protocol) — Bedside ultrasound will be used to view any intraperitoneal bleeding, pleural fluid, cardiac abnormalities, or structural abnormalities of major blood vessels. The results of this test will then be used to determine the best course of treatment for the patient.
  Arms: Ultrasound

SUMMARY:
This study is designed to determine if there is any relationship between performing an abdominal ultrasound on patients who present with hypotension and their clinical outcomes (as measured by 7, 30 day and discharge mortality).

DETAILED DESCRIPTION:
STRUCTURED RESEARCH ABSTRACT

Introduction

Patients who present to the ED (emergency department) with undifferentiated, non-trauma associated hypotension are often affected by conditions with a prognosis largely dependent on the time taken from presentation to correct diagnosis and intervention. The ACES protocol (Abdominal and Cardiothoracic Evaluation with Sonography in Shock) provides a rapid focused ultrasound protocol for making or refining diagnoses in patients who present to the ED with this type of hypotension. This will be the first study to compare the clinical outcomes of patients who are assessed with the ACES protocol as part of their initial workup to those of patients who are assessed without any intervention by ultrasound. The goal of this study is to determine if ACES enhances the patient's clinical outcomes, as measured by: 1) Time to restoration (or improvement) of CVS (cardiovascular system) parameters, 2) Rate of normalization of acid-base balance, as well as venous lactate 3) Significant change in diagnosis or recommended intervention 4) Frequency of unexpected diagnosis, and 5) Patient 7 and 30-day, and discharge mortality rate.

Methods

SHoC-ED 1 is a stratified randomized control trial that will run in multiple centers across Canada and internationally. The data will be stratified in that each center involved will recruit equal amounts of control and intervention patients. While different centers will recruit different numbers of participants, each individual center will recruit near-equal amounts for each arm of the study.

ED nurses will identify potential candidates for the SHoC-ED 1 study, and flag their charts to notify the attending physician. ED Physicians trained on the ACES protocol will then proceed to review the exclusion criteria (part of patient inclusion sheet/patient flag) and where appropriate, obtain consent. After these are completed, the physician will retrieve an envelope that contains the already randomized forms appropriate for whichever arm the patient has been randomized to. This randomization will place patients in either the ACES group (to be referred to as Group 1), or the control group (to be referred to as Group 2). Physicians following the group 1 protocol will perform their normal initial assessment and then do ACES, recording their data after each step. Physicians in group 2 will simply record their data after the initial assessment. Both groups of physicians will then record their impressions at 60 minutes as this will enable this project to determine how changes in diagnoses are affected by non-ultrasound factors in the first hour a patient is in the ED. These diagnoses will then be compared against the "final" diagnoses made during the patient's admission. Exclusion criteria for this study include the following: A) necessity of CPR or other advanced life support interventions before enrollment, B) History of significant trauma in past 24 hours, C) A 12 lead ECG diagnostic of STEMI, D) Mechanism of shock is clear (i.e. not undifferentiated shock), E) previously known diagnosis from other hospital, F) previously confirmed pregnancy, G) vagal episode H) Low blood pressure is not actually pathologic hypotension, but instead a normal variant or some other phenomenon.

To ensure that scans are being performed properly and consistently at all sites included in this study local principal investigators will be responsible for ensuring appropriate training and monitoring of standards for the physicians at their center performing ACES.

The data collected from both Group 1 and Group 2 will then be compared against each other, and follow-up will be conducted to ascertain if the early intervention with ACES had any implications on long-term outcomes.

Results

Given that much of the data interpreted will be comparing numerical values from different strata (Example: Time taken to operating theatre compared between Group 1 and 2), ANOVA testing will be used. The results of the ANOVA test will be used to determine if there is a significant difference in outcome, as measured by 1) Time to restoration (or improvement) of CVS parameters, and 2) Rate of normalization of acid-base balance (using either venous or arterial blood gas), and blood lactate.

For categorical data (Example: Mortality rate between groups), chi-square analyses will be performed to determine statistically significant increase in clinical outcome. This will be done for:

* Significant changes in diagnosis/recommendations in intervention change, and
* Frequency of unexpected diagnosis.

Conclusion

This SRCT (stratified randomized control trial) will determine whether the ACES protocol leads to improved clinical outcomes in patients who present to the ED with undifferentiated, non-trauma associated shock. It will compare intervention with the ACES protocol to intervention with no ultrasound at all.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Systolic Blood Pressure under 100 OR Systolic BP under pulse (up to 120)

Exclusion Criteria:

* Patients known to be pregnant at time of presentation
* Necessity of CPR or other advanced life support interventions before enrolment
* History of significant trauma in past 24 hours
* A 12 lead diagnostic of acute myocardial infarction
* Mechanism of shock is clear (i.e. not undifferentiated shock)
* Previously known diagnosis from other hospital
* Vagal episode (as cause of hypotension)
* Low blood pressure not actually being pathologic hypotension (Normal Variant or other)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Patient Mortality Rates (7-day, 30 Day or Hospital Discharge) | 7-day, 30 Day or Hospital Discharge
  Determine the proportion of patients living at 7-day, 30 Day or Hospital Discharge

SECONDARY OUTCOMES:
Time taken to appropriate intervention | Within 8 hours
  This is a measure that will be done to determine how long after initial diagnosis "appropriate" interventions are taken. This will be done by reviewing the patient's chart, identifying what the ultimate diagnosis for the patient was (resultant of testing that occurs as patient progresses through system), and seeing when propoer intervention was taken.
Unexpected change in diagnosis | First hour
  If ED physician's expectations prior to performing ultrasound is AAA, but post ultrasound diagnosis is septic shock, this would be an example of an unexpected change in diagnosis. This measure will only be performed in the ultrasound group, as the purpose is to identify how often performing ultrasound will result in diagnosis changes.

CONTACTS AND LOCATIONS:
Overall Officials: James D Milne, MD (Student), Principal Investigator — Dalhousie Medical School; Paul Atkinson, MD, Principal Investigator — Saint John Regional Hospital, Horizon Health Network; Jacqueline Fraser, BN, Study Director — Saint John Regional Hospital, Horizon Health Network
Locations (6):
- Canada (3):
  - University of Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Saskatoon Health Region, Saskatoon, Saskatchewan
- South Africa (3):
  - GF Jooste Hospital, Manenberg, Cape Town
  - Tygerberg Hospital, Cape Town, Western Cape
  - Khayelitsha Hospital, Cape Town

REFERENCES:
- [Result] Atkinson PR, Milne J, Diegelmann L, Lamprecht H, Stander M, Lussier D, Pham C, Henneberry R, Fraser JM, Howlett MK, Mekwan J, Ramrattan B, Middleton J, van Hoving DJ, Peach M, Taylor L, Dahn T, Hurley S, MacSween K, Richardson LR, Stoica G, Hunter S, Olszynski PA, Lewis DA. Does Point-of-Care Ultrasonography Improve Clinical Outcomes in Emergency Department Patients With Undifferentiated Hypotension? An International Randomized Controlled Trial From the SHoC-ED Investigators. Ann Emerg Med. 2018 Oct;72(4):478-489. doi: 10.1016/j.annemergmed.2018.04.002. Epub 2018 Jun 2. PMID 29866583